CLINICAL TRIAL: NCT01331837
Title: A Clinical Outcomes Study to Evaluate the Effects of IL-6 Receptor Blockade With Tocilizumab (TCZ) in Comparison With Etanercept (ETA) on the Rate of Cardiovascular Events in Patients With Moderate to Severe Rheumatoid Arthritis (RA)
Brief Title: A Study of Tocilizumab in Comparison to Etanercept in Participants With Rheumatoid Arthritis and Cardiovascular Disease Risk Factors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WA25204; 2010-020065-24 (EudraCT Number)
Record Dates: First submitted 2011-04-07; First posted 2011-04-08 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; tocilizumab

ARMS (2):
- Etanercept (Active Comparator)
  Interventions: Drug: Etanercept
- Tocilizumab (Experimental)
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Etanercept — Participants will receive 50 mg etanercept subcutaneously weekly until switch to another RA therapy or up to 4.9 years.
  Arms: Etanercept
Drug: Tocilizumab — Participants will receive 8 mg/kg tocilizumab IV every 4 weeks until switch to another RA therapy or up to 4.9 years.
  Other Names: Actemra
  Arms: Tocilizumab

SUMMARY:
This randomized, open-label, parallel-group, multicenter study will evaluate the rate of cardiovascular events with tocilizumab in comparison to etanercept in participants with rheumatoid arthritis (RA). Participants will be randomized to receive intravenous (IV) 8 milligrams per kilogram (mg/kg) tocilizumab every 4 weeks or subcutaneous 50 milligrams (mg) etanercept weekly, with or without non-biologic disease-modifying anti-rheumatic drug (DMARD).

ELIGIBILITY:
Inclusion Criteria:

* Participants with moderate to severe RA of greater than or equal to (>=6) months duration
* Inadequate response to at least one non-biologic DMARD
* Positive for Rheumatoid Factor (RF) and/or anti-cyclic citrullinated peptide (CCP) antibodies at screening
* Have C-reactive protein (CRP) greater than (>) 0.3 milligrams per deciliter (mg/dL) at screening or at the baseline visit
* Swollen joint count (SJC) >=8 (66 joint count) and tender joint count (TJC) >= 8 (68 joint count) during screening or at the baseline visit
* History of Coronary Heart Disease (CHD) or presence of one or more additional CHD risk factors, including current cigarette smoking, hypertension, low High Density Lipoprotein (HDL) cholesterol, family history of premature CHD, diabetes, presence of extra-articular disease associated with rheumatoid arthritis
* At the time of randomization, will have discontinued infliximab, adalimumab, golimumab, or certolizumab for >= 4 weeks

Exclusion Criteria:

* Major surgery (including joint surgery or coronary revascularization) within 8 weeks prior to screening or planned major surgery within 1 year of study start
* Rheumatic autoimmune disease other than RA
* History of or current inflammatory joint disease other than RA
* Current or recent (within past 3 months) evidence of serious uncontrolled concomitant cardiovascular or cerebrovascular disease (myocardial infarction, revascularization, stroke, transient ischemic attack, or acute coronary syndrome)
* Current or previous (within the past 2 years) evidence of serious uncontrolled concomitant pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (including uncontrolled diabetes mellitus) or gastrointestinal disease
* Uncontrolled disease states, such as asthma or inflammatory bowel disease where flares are commonly treated with oral or parenteral corticosteroids
* Pre-existing central nervous system demyelinating or seizure disorders
* History of diverticulitis, diverticulosis requiring treatment or other lower gastrointestinal tract conditions that might predispose to perforations
* Current liver disease as determined by the investigator; a history of asymptomatic elevations in liver function tests (LFTs) is not considered an exclusion
* Active current infection or history of recurrent bacterial, viral, fungal, mycobacterial or other infections, including but not limited to tuberculosis and atypical mycobacterial disease, hepatitis B and C, and herpes zoster, but excluding fungal infections of nail beds
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within four weeks of screening or oral antibiotics within two weeks prior to screening visit
* Active tuberculosis (TB) requiring treatment within 3 years prior to baseline
* Latent TB diagnosed during screening that has not been appropriately treated
* Primary or secondary immunodeficiency (history of or currently active)
* Moderate to severe heart failure
* Evidence of active malignant disease, malignancies diagnosed within the previous 10 years (including hematologic malignancies and solid tumors, except basal cell carcinoma of the skin that has been excised and cured), or breast cancer diagnosed within the previous 20 years
* Breast feeding mothers
* History of alcohol, drug or chemical abuse within the 6 months prior to screening
* Participants with lack of peripheral venous access
* Participants with a history of allergic reactions to latex
* Previous treatment with non-tumor necrosis factor (non-TNF)-inhibitor biologic therapy
* Treatment with any investigational agent within 4 weeks of screening visit
* Treatment with any cell depleting therapies within 1 year of baseline
* Treatment with IV gamma globulin, plasmapheresis or Prosorba column within 6 months of baseline visit
* Immunization with a live/attenuated vaccine within 4 weeks prior to baseline visit
* Any previous treatment with alkylating agents, such as cyclophosphamide or chlorambucil, or with total lymphoid irradiation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3080 (Actual)
Dates: Start 2011-08-02 (Actual); Primary Completion 2016-03-25 (Actual); Study Completion 2016-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (428):
- United States (143):
  - Uni Of Alabama,Birmingham; Medicine - Rheumatology, Birmingham, Alabama
  - Rheumatology Associates of North Alabama, Huntsville, Alabama
  - Clinical and Translational Research Center of Alabama, PC, Tuscaloosa, Alabama
  - Arizona Arthritis & Rheumatology Associates, P.C., Glendale, Arizona
  - Arizona Arthritis & Rheumatology Research, Pllc, Paradise Valley, Arizona
  - Sun Valley Arthritis Center, Peoria, Arizona
  - Valley Arthritis Care, Phoenix, Arizona
  - Advanced Arthritis Care & Research, Scottsdale, Arizona
  - Camp Lowell Medical Specialists, Tucson, Arizona
  - The University of Arizona, Tucson, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - OrthoArkansas; Orthopedics & Sports Medicine, Little Rock, Arkansas
  - Samy Metyas, MD, Inc, Covina, California
  - Talbert Medical Group, Huntington Beach, California
  - Allergy & Rheumatology Medical Clinic, Inc, La Jolla, California
  - Valerius Medical Group, Los Alamitos, California
  - Clinical Interventions Research Institute, Mission Viejo, California
  - Dr. Brigid Freyne, MD, Murrieta, California
  - Sharp Rees-Stealy Medical Group, Poway, California
  - San Diego Arthritis Med Clnc, San Diego, California
  - Purushotham & Akther Kotha Inc, San Diego, California
  - C Michael Neuwelt MD Inc, San Leandro, California
  - Pacific Arthritis Ctr Med Grp, Santa Maria, California
  - Orrin M. Troum, Md, Santa Monica, California
  - Harbor UCLA Medical Center, Torrance, California
  - Inland Rheumatology; Clinical Trials, Inc., Upland, California
  - Medvin Clinical Research, Whittier, California
  - Arthritis Assoc & Osteoporosis; Ctr of Colorado Springs, Colorado Springs, Colorado
  - Joao Nascimento, Bridgeport, Connecticut
  - University of Connecticut Health Center, Farmington, Connecticut
  - Arthritis & Osteoporosis Center Pc, Hamden, Connecticut
  - ZASA Clinical Research, Boynton Beach, Florida
  - DC Health Clinic, Coral Gables, Florida
  - Tsai, Yong, Daytona Beach, Florida
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - Pharmax Research Clinic Inc., Miami, Florida
  - Arthritis/Osteoporosis Treatment Center, Orange Park, Florida
  - Arthritis Rsrch of Florida, Inc., Palm Harbor, Florida
  - Baptist Hospital Clinical Research, Pensacola, Florida
  - Lovelace Scientific Resources, Sarasota, Florida
  - Centre for Arthritis and Rheumatic Diseases, South Miami, Florida
  - Pinellas Medical Research, LLC, St. Petersburg, Florida
  - SW Florida Clinical Research, Tampa, Florida
  - Healthpoint Medical group, Inc, Tampa, Florida
  - Emory Uni ; Division of Rheumatology, Atlanta, Georgia
  - Arthritis & Rheumatology of Georgia, Atlanta, Georgia
  - North Georgia Rheumatology, Duluth, Georgia
  - Harbin Clinic, Rome, Georgia
  - St. Joseph'S/Candler Health System, Inc.; Office of Research, Savannah, Georgia
  - Sonora Clinical Research, Boise, Idaho
  - St. Luke's Intermountain Research Center, Boise, Idaho
  - Selah Medical Ctr, Boise, Idaho
  - Coeur D'Alene Arthritis Clinic, Coeur d'Alene, Idaho
  - Idaho Arthritis Center, Meridian, Idaho
  - University of Illinois at Chicago, Chicago, Illinois
  - Apex Medical Research, AMR, Inc., Chicago, Illinois
  - Methodist Medical Center of Ilinois, Peoria, Illinois
  - Northern Indiana Research Alliance, Fort Wayne, Indiana
  - Diagnostic Rheumatology & Research, Indianapolis, Indiana
  - Memorial Medical Group Clinical Research, South Bend, Indiana
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Research Integrity, Owensboro, Kentucky
  - Arthritis & Diabetes Clinic, Inc, Monroe, Louisiana
  - Ochsner Health System, New Orleans, Louisiana
  - Rheumatology Associates of Baltimore, Baltimore, Maryland
  - Osteoporosis & Clinical Trials Center, Hagerstown, Maryland
  - Center For Rheumatology & Bone Research, Wheaton, Maryland
  - Phase Iii Clinical Research, Fall River, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Hurley Research Center, Flint, Michigan
  - Rheumatology, P.C.; Medical Arts Building, Kalamazoo, Michigan
  - Advanced Rheumatology, PC, Lansing, Michigan
  - Northern Michigan Regional Hospital, Petoskey, Michigan
  - St. Paul Rheumatology, Eagan, Minnesota
  - Va Medical Center, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Jackson Arthritis Clinic, Flowood, Mississippi
  - North Mississippi Med Clinics, Inc., Tupelo, Mississippi
  - Glacier View Research Institute, Kalispell, Montana
  - Univ of Nebraska Medical Ctr, Omaha, Nebraska
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Innovative Health Research, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Rheumatology 5C, Lebanon, New Hampshire
  - Nashua Rheumatology - Foundation Medical Partners, Nashua, New Hampshire
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Rheumatology Associates Of New Jersey, Teaneck, New Jersey
  - Arthritis Rheumatic & Back Disease Associates, Voorhees Township, New Jersey
  - Albuquerque Center For Rheumatology, Albuquerque, New Mexico
  - Arthritis and Osteoporosis Associates of New Mexico, Las Cruces, New Mexico
  - Arthritis & Osteoporosis Medical Associates, Pllc, Brooklyn, New York
  - SUNY Downstate Medical Center., Brooklyn, New York
  - DiGiovanna Inst for Med Ed&Res, North Massapequa, New York
  - Southern Tier Arthritis & Rheumatism, Olean, New York
  - Arthritis Health Associates; Clinical Research, Syracuse, New York
  - Asheville Arthritis & Osteoporosis Center, PA, Asheville, North Carolina
  - Joint & Muscle Research Institute, Charlotte, North Carolina
  - Carolina Bone & Joint P.A., Charlotte, North Carolina
  - Durham Rheumatology, Durham, North Carolina
  - PMG Research of Hickory LLC, Hickory, North Carolina
  - Shanahan Rheumatology & Immunology, PLLC, Raleigh, North Carolina
  - Specialty Medical Clinic and Research Center, Sanford, North Carolina
  - Carolina Arthritis Associates, Pa, Wilmington, North Carolina
  - Trinity Health Center, Minot, North Dakota
  - Cincinnati Rheumatic Disease Study Group, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Ohio State Univ Med Center, Columbus, Ohio
  - Columbus Arthritis Center, Columbus, Ohio
  - Clinical Research Source, Inc., Toledo, Ohio
  - Toledo Clinic, Toledo, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Ilumina Clinical Associates, Indiana, Pennsylvania
  - PMA Medical Specialists, Limerick, Pennsylvania
  - Pivotal Clinical Research, Llc, Perkasie, Pennsylvania
  - Arthritis Group, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Health System; Infectious Disease, Pittsburgh, Pennsylvania
  - Allegheny Rheumatology, Wexford, Pennsylvania
  - Clinical Research Center of Reading, Wyomissing, Pennsylvania
  - Pennsylvania Regional Center for Arthritis and Osteoporosis Research, Wyomissing, Pennsylvania
  - Columbia Arthritis Center (Partnership Practice), Columbia, South Carolina
  - South Carolina Research Center, Myrtle Beach, South Carolina
  - Brown Clinic, Watertown, South Dakota
  - Ramesh Gupta - PP, Memphis, Tennessee
  - Amarillo Center For Clinical Research, Amarillo, Texas
  - Adriana Pop-Moody MD Clinic PA, Corpus Christi, Texas
  - Metroplex Clinical Research, Dallas, Texas
  - Leading Edge Research, PA; Office of Dr. Burbano, Fort Worth, Texas
  - Rheumatic Disease Clin Res Ctr, Houston, Texas
  - Houston Inst. For Clinical Research, Houston, Texas
  - Southwest Rheumatology, Mesquite, Texas
  - Leading Edge Research, PA; Office of Dr. Burbano, Richardson, Texas
  - Texas Arthritis Research Center, San Antonio, Texas
  - Arthritis & Osteoporosis Clinic, Waco, Texas
  - Arthritis and Rheumatic Disease Associates, Burke, Virginia
  - Sentara Medical Group, Norfolk, Virginia
  - Apex Clinical Research, Kennewick, Washington
  - Seattle Rheumatology Associates, Seattle, Washington
  - Office of George Krick, Md, Tacoma, Washington
  - Rheum & Pulmonary Clinic, Beckley, West Virginia
  - Mountain State Clinical Research, Clarksburg, West Virginia
  - Arthritis Centre; Suite 103, Racine, Wisconsin
- Argentina (21):
  - Centro de Investigaciones Reumatologicas y Osteologicas, Buenos Aires
  - Organizacion Medica de Investigacion, Buenos Aires
  - CEIM Consultorios Especializados en Investigaciones Médicas, Buenos Aires
  - APRILLUS, Buenos Aires
  - Instituto centenario, Buenos Aires
  - Fundación CIDEA, Buenos Aires
  - Atencion Integral En Reumatologia Buenos Aires, Buenos Aires
  - CEMIC, Buenos Aires
  - Hospital General de Agudos Dr. J. M. Ramos Mejia, Ciudad Autonoma Buenos Aires
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Hospital Privado Cordoba, Cordoba Pcia
  - Instituto Reumatológico Strusberg, Córdoba
  - Hospital Italiano de Cordoba, Córdoba
  - Hospital Municipal Nuestra Sra. de Lujan, Luján
  - Centro de Investigacion Pergamino SA, Pergamino
  - Sanatorio Parque de Rosario, Rosario
  - Instituto Centralizado de Asistencia e Investigaci, Rosario, Santa Fe
  - CER San Juan Centro Polivalente de Asistencia e Investigacion Clinica, San Juan
  - Centro de Investigaciones Médicas - CIM, San Juan Bautista
  - Centro de Investigaciones Reumatologicas Tucuman, San Miguel de Tucumán
  - Centro Médico Privado de Reumatología, San Miguel de Tucumán
- Austria (5):
  - Lkh-Univ. Klinikum Graz, Graz
  - Landesklinikum Weinviertel Stockerau; Rheumatologie, Stockerau
  - Medizinische Universität Wien, Vienna
  - Rheuma-Zentrum Favoriten Wien, Vienna
  - Krankenhaus Hietzing; 2.Med.Abteilung, Pav.3A, Vienna
- Belgium (5):
  - CHU St Pierre (St Pierre), Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - AZ Groeninge (Vercruysselaan), Kortrijk
  - CHU Sart-Tilman, Liège
  - ZNA Jan Palfijn, Merksem
- Bosnia and Herzegovina (4):
  - University Clinical Center of the Republic of Srpska, Banja Luka
  - University Clinic Ctr Sarajevo, Sarajevo
  - General Hospital Prim.dr.Abdulah Nakas, Sarajevo
  - Uni Hospital Center Tuzla, Tuzla
- Canada (17):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - The Medical Arts Health Research Group, Powell River, British Columbia
  - Baker, Milton F., Victoria, British Columbia
  - Nexus Clinical Research Centre, St. John's, Newfoundland and Labrador
  - St. Clare'S Mercy Hospital, St. John's, Newfoundland and Labrador
  - Arthur Karasik, MD, Etobicoke, Ontario
  - Charlton Medical Center, Hamilton, Ontario
  - K-W Musculoskeletal Research, Kitchener, Ontario
  - St. Joseph's Hospital, London, Ontario
  - Credit Valley, Rheumatology, Mississauga, Ontario
  - Niagara Peninsula Arthritis Centre, St. Catharines, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Institut de Rhumatologie de Montreal, Montreal, Quebec
  - Groupe de Recherche En Rhumatologie Et Maladies Osseuses, Québec, Quebec
  - Chus Hopital Fleurimont, Sherbrooke, Quebec
  - Centre de Recherche Musculo-Squelettique, Trois-Rivières, Quebec
  - Centre Re Recherche Saint-Louis, Québec
- Chile (9):
  - Hospital San Juan de Dios La Serena, La Serena
  - Centro Medico Prosalud, Santiago
  - Interin, Santiago
  - Centro de Estudios Reumatológicos, Santiago
  - Hospital Clinico Pontificia Universidad Catolica de Chile, Santiago
  - Centro de Investigacion Clinica del Sur, Temuco
  - Clinica Alemana de Temuco, Temuco
  - Hospital Clinico Viña del Mar- Oncovida, Viña del Mar
  - Centro de Estudios Clinicos V Region Limitada, Viña del Mar
- Croatia (5):
  - General Hospital Karlovac, Karlovac
  - Special Hospital for Medical Rehabilitation, Krapinske Toplice
  - Clinical Hospital Centre Rijeka; Department of Rheumatology and Clinical Immunology, Rijeka
  - Clinical Hospital Centre Zagreb, Zagreb
  - Universtiy Hospital Dubrava, Zagreb
- Czechia (12):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Revmatologicka ambulance, Bruntál
  - Revmatologicka Ambulance, Hlučín
  - Interni a revmatologicka ordinace, Hostivice
  - Revmatologicka a-interni ambulance, Kladno
  - Revmatologie MUDr. Klara Sirova s.r.o., Ostrava - Moravska Ostrava
  - Revmatologicky Ustav, Prague
  - Revmatologicka ambulance, Prague
  - Fakultni Thomayerova nemocnice s poliklinikou, Prague
  - Artroscan s.r.o., Sokolov
  - Revmatologicka Ambulance-Terezin, Terezín
  - PV - Medical, s.r.o., Zlín
- Ecuador (6):
  - Hospital Clínica Santa Inés, Cuenca
  - Centro de Reumatología y Rehabilitación, Guayaquil
  - OMNI Hospital, Guayaquil
  - Centro Medico Alcivar 4, Guayaquil
  - Centro Medico Picasso, Quito
  - Novaclinica Santa Cecilia; Reumatology, Quito
- France (16):
  - CHU d'Amiens Hôpital Nord; Pharmacie Clinique, Amiens
  - Groupe Hospitalier Pellegrin, Bordeaux
  - CHU Hopital Gabriel Montpied, Clermont-Ferrand
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CHU Grenoble Sud, Échirolles
  - Hôpital Edouard Herriot; Service de Rhumatologie, Lyon
  - CHR Orleans, Hopital Madeleine, Orléans
  - Hôpital Saint-Antoine; Service de Psychiatrie, Paris
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - Hopital Cochin; Gastro Enterologie, Paris
  - Hôpital Sud - CHU de Rennes, Rennes
  - Hôpital Victor Provo, Roubaix
  - CHU de Rouen, Hopital de Bois Guillaume; Service de Rhumatologie, Rouen
  - CHU Saint-Etienne, Hopital Bellevue, Saint-Etienne
  - Hôpital General - CHRU de Dijon, Strasbourg
  - Institut Universitaire du Cancer - Oncopole Toulouse (IUCT-O), Toulouse
- Germany (16):
  - Charité Universitaetsmedizin Berlin, Campus Charité Mitte, Berlin
  - Schlosspark-Klinik, Berlin
  - Universitätsklinikum Köln, Klinik I für Innere Medizin, Cologne
  - Universitätsklinikum "Carl Gustav Carus" der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Erlangen; Augenklinik, Erlangen
  - Praxisgemeinschaft Rheumatologie-Nephrologie Erlangen PGRN, Erlangen
  - Universitaetsklinikum Frankfurt, Frankfurt
  - Universitaetsklinikum Hamburg-Eppendorf; Medizinische Klinik Nephrologie/Rheumatologie, Hamburg
  - Schön Klinik Hamburg-Eilbek Klinik für Rheumatologie, Hamburg
  - Rheumazentrum Ruhrgebiet; St. Josefs-Krankenhaus, Herne
  - Gemeinschaftspraxis Dr. Von Hinueber/Dr. Demary; Rheumatologie, Hildesheim
  - Universitaetsklinikum Leipzig, Leipzig
  - Ludwig Maximilians; Universitaet, München
  - Praxiszentrum St. Bonifatius, München
  - Rheumatologische Gemeinschaftspraxis, Osnabrück
  - Evangelisches Fachkrankenhaus, Ratingen
- Greece (7):
  - Laiko General Hospital Athen, Athens
  - Euroclinic of Athens; Internal Medicine & Immunology Dept., Athens
  - University General Hospital of Heraklion, Crete
  - University General Hospital of Larissa; Rheumatology Unit, Larissa
  - General Hospital of Thessaloniki Hippokration, Thessaloniki
  - Euromedica Kyanous Stavros General Hospital, Thessaloniki
  - 424 Military Training Hospital-Egnatia, Thessaloniki
- Hungary (11):
  - Országos Fizioterápiás És Reumatológiai Intézet; I. Reumatológiai És Metabolikus Osteológiai Osztály, Budapest
  - Clinexpert Egeszsegugyi Szolgaltato es Kereskedelmi Kft, Budapest
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Synexus Magyarorszag Kft, Budapest
  - Debreceni Egyetem, Klinikai Kozpont, Tudogyogyaszati Klinika, Debrecen
  - Markhot Ferenc Eu. Szolg. Nonprofit Kiem. Kozh. Kft., Eger
  - Bekes Megyei Kepviselotestulet Pandy Kalman Korhaza, Gyula
  - Varosi Korhaz-Rendelointezet, Mór
  - Clinfan Szolgaltato Kft., Szekszárd
  - Fejer Megyei Szent Gyorgy Korhaz, Székesfehérvár
  - Zala Megyei Korhaz; Reumatologia, Zalaegerszeg
- India (7):
  - Shalby Hospital Limited, Ahmedabad, Gujarat
  - Vedanta Institute; Medical Sciences, Ahmedabad
  - Manipal Hospital, Bangalore
  - St.John's Medical College Hospital, Banglore
  - Arthritis Super Speciality Centre, Hubli
  - Care Institute of Medical Sciences, Hyderabad
  - Jasleen Hospital, Nagpur
- Israel (5):
  - Barzilai Medical Center, Ashkelon
  - Assaf Harofeh Medical Center, Beer Yaacov
  - The Lady Davis Carmel Medical Center, Haifa
  - Chaim Sheba Medical Center; Rheumatology, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (11):
  - Azienda Ospedaliera A. Cardarelli, Napoli, Campania
  - Ospedale San Giovanni Bosco; Divisione di Reumatologia, Napoli, Campania
  - Fondazione Salvatore Maugeri IRCCS; Istituto Scientifico di Riabilitazione di Telese, Telese Terme, Campania
  - Ospedale La Colletta, Arenzano, Liguria
  - Azienda Ospedaliero Universitaria San Martino, Genoa, Liguria
  - Ospedali Riuniti di Bergamo, Bergamo, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - Ospedale Di Circolo E Fondazione Macchi, Varese, Lombardy
  - Presidio Ospedaliero Vittorio Emanuele, Catania, Sicily
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Ospedale Misericordia e Dolce, Prato, Tuscany
- Latvia (7):
  - L.Krumina GP practice, Bauska
  - Daugavpils Regional Hospital, Daugavpils
  - D.Saulite-Kandevica Private Practice, Liepāja
  - Clinic ORTO, Riga
  - Private Practice EHOKG, Riga
  - Riga East Clinical University Hospital; Clinic Gailezers, Riga
  - P. Stradins Clinical University Hospital, Riga
- Lithuania (5):
  - Alytus Regional S. Kudirkos Hospital, Public Institution, Alytus
  - Klaipeda Seamen's Hospital, Public Institution, Klaipėda
  - Klaipeda University Hospital; Public Institution, Klaipėda
  - Siauliai Republican Hospital Public Institution, Šiauliai
  - Vilnius District Central Outpatient Clinic, Public Institution, Vilnius
- Malaysia (6):
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Sunway Medical Centre, Kuala Selangor, Selangor
  - Sime Darby Medical Centre, Kuala Selangor, Selangor
  - Hospital Selayang, Kuala Lumpur
  - Hospital Umum Sarawak, Kuching
- Mexico (23):
  - Centro de Investigacion del Noroeste SC, Tijuana, Estado de Baja California
  - Centro de Investigación de Tratamientos Innovadores de Sinaloa (CITI), Culiacán, Sinaloa
  - Unidad de Atencion Medica e Investigacion en Salud S.C., Mérida, Yucatán
  - Hospital Christus Muguerza del Parque; Reumatologia, Chihuahua City
  - Hospital CIMA Chihuahua; Reumatologia, Chihuahua City
  - Hospital Privado San Jose de Ciudad Obregon SA de CV, Ciudad Obregón
  - Private Practice Dr. Cortes, Cuernavaca
  - RM pharma specialist SA de CV, Delegacion Benito Juarez
  - Mentrials S.A. de C.V, Distrito Federal
  - Centro de Investigacion y Atencion Integral Durango CIAID, Durango
  - Mundo Fisico, Guadalajara
  - Clinica Hospital Angeles Chapalita, Guadalajara
  - Centro de Investigacion en Enfermedades Reumaticas y Osteoporosis, Mexicali
  - Inst. Mexicano de Investigacion Clinica, Mexico City
  - Hospital Mocel, Mexico City
  - Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City
  - Mexico Centre for Clinical Research, México
  - Comite Mexicano Para la Prevencion de Osteoporosis AC, México
  - Cliditer SA de CV, Miexico City
  - Hospital Universitario de Saltillo, Saltillo
  - Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosi S.l.p.
  - Centro de Alta Especialidad en Reumatología e Investigación del Potosí, S.C., San Luis Potosí City
  - Unidad de Enfermedades Reumaticas y Cronicodegenerativas, Torreón
- Netherlands (4):
  - Jan Van Breemen Instituut, Amsterdam
  - Albert Schweitzer Ziekenhuis ; Dordwijk, Dordrecht
  - Franciscus Ziekenhuis, Roosendaal
  - Vlietland Hospital, Schiedam
- Philippines (5):
  - Cebu Doctors' University Hospital- North General Hospital, Cebu City
  - Chong Hua Hospital, Cebu City, Cebu City
  - St. Paul Hospital; Arthritis Center, Iloilo City
  - Mary Mediatrix Medical Center, Lipa City
  - Makati Medical Center, Makati City
- Poland (11):
  - Szpital Uniwersytecki; nr 2 im. Dr J. Biziela, Bydgoszcz
  - Wojewodzki Szpital Zespolony w Elblagu, Elblag
  - Szpital Specjalistyczny Im J. Dietla Malopolskie Centrum Reumat; Oddzial Rumatologii, Krakow
  - Szpital Specjalistyczny im. J. Dietla, Krakow
  - NZOZ REUMED Sp. z o.o., Lublin
  - Lecznica MAK-MED NZOZ, Nadarzyn
  - SP Szpital Kliniczny nr 1 Pomorskiej Akademii Medycznej im. prof. Tadeusza Sokolowskiego, Szczecin
  - Slaski Szpital Reumatologiczno; Rehabilitacyjny; Iii Oddzial Reumatologiczny, Ustroń
  - Rheuma Medicus Zaklad Opieki Zdrowotnej, Warsaw
  - ARS Rheumatica Sp.z o. o, Warsaw
  - Akademicki Szpital Kliniczny im. Jana Mikulicza Radeckiego, Wroclaw
- Romania (13):
  - Spitalul Clinic Judetean de Urgenta Brasov, Brasov
  - Spitalul Clinic Sf. Maria; Dept Interna si Reumatologie, Bucharest
  - Spitalul Clinic Dr. I Cantacuzino, Bucharest
  - Centrul de Boli Reumatismale Dr. Ioan Stoia, Bucharest
  - Medex SRL, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Clinica de Medicina Muncii, Cluj-Napoca
  - CMI Dr.Ciornohuz Adriana, Iași
  - Spitalul Clinic de Recuperare Iasi, Iași
  - Spitalul Municipal Ploiesti, Ploieşti
  - Spitalul Clinic Colentina, Sector 2
  - Spitalul Judetean de Urgenta Targoviste, Târgovişte
  - Mediab SRL, Târgu Mureş
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara
- Russia (17):
  - State institution of health care - Territorial Clinical Hospital, Barnaul
  - SEI of HPE "Altay State Medical University of Roszdrav", Barnaul
  - Scientific and research medical complex Your Health, Kazan'
  - SIH Kemerovo Regional Clinical Hospital, Kemerovo
  - City Hospital No.4, Moscow
  - Scient Res Inst Rheumat RAMS, Moscow
  - Moscow State Medical Stomatological University, Moscow
  - Head Clinical Hospital of Internal Affair Ministry of Russia, Moscow
  - MHI City Clinical Hospital#19, Novosibirsk
  - FSBI Scientific Research Institute of Clinical Immunology of SB of RAMS, Novosibirsk
  - Ryazan Regional Clinincal Cardiology Dispensary, Ryazan
  - Leningradskaya Regional Clinical Hospital; Rheumatology Dept, Saint Petersburg
  - State institution of healthcare "Regional hospital for war veterans", Saratov
  - Stavropol State Medical Academy, Stavropol
  - Tomsk Regional Clinical Hospital, Tomsk
  - Voronezh Regional Clinical Hospital #1, Voronezh
  - MCHI Medical Sanitary Unit of Yaroslavl Diesel Apparatus Plant, Yaroslavl
- Serbia (4):
  - Institute of Rheumatology, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Bezanijska Kosa, Belgrade
  - Institute of Rheumatology and Cardiovascular Diseases; Rheumatology, Niška Banja
- South Africa (4):
  - Groote Schuur Hospital; Rheumatology Unit, Cape Town
  - Chris Hani Baragwanath Hospital; Rheumatology Department, Diepkloof
  - Charlotte Maxeke Academic Hospital, Johannesburg
  - University of Pretoria; Clinical Trial Unit, Pretoria
- Spain (12):
  - Hospital de Merida ;Servicio de Reumatologia, Mérida, Badajoz
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Sierrallana, Torrelavega, Cantabria
  - Hospital General de Castellon; Servicio de Reumatologia, Castellon, Castellon
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital Infanta Sofia; Servicio de Reumatologia, San Sebastián de los Reyes, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga, Malaga
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital Universitario de Canarias, S. Cristobal de La Laguna, Tenerife
  - Hospital de Cruces; Servicio de Reumatologia, Barakaldo, Vizcaya
  - Hospital Universitario Basurto, Bilbao, Vizcaya
  - Hospital Gregorio Marañon, Madrid
- Turkey (Türkiye) (4):
  - Akdeniz Univesity Medical Faculty, Antalya
  - Trakya University Medical Faculty, Edirne
  - Ataturk University Med Faculty, Erzurum
  - Karadeniz Tecnical Uni. Med. Fac., Trabzon
- United Kingdom (13):
  - Selly Oak Hospital; Rheumatology Dept, Birmingham
  - Addenbrooke's NHS Trust, Cambridge
  - Cannock Chase Hospital; Rheumatology, Cannock
  - Russells Hall Hospital; Rheumatology Department, Dudley
  - Leicester Royal Infirmary NHS Trust, Leicester
  - Royal London Hospital Outpatients Department, London
  - Whipps Cross Hospital; Rheumatology Dept, London
  - King'S College Hospital, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Salford Royal NHS Foundation Trust, Salford
  - Southampton General Hospital; Rheumatology, Southampton
  - Southend Hospital; Rheumatology Department, Westcliffe-on-sea
  - Wrightington Hospital, Wrightington

REFERENCES:
- [Derived] Giles JT, Sattar N, Gabriel S, Ridker PM, Gay S, Warne C, Musselman D, Brockwell L, Shittu E, Klearman M, Fleming TR. Cardiovascular Safety of Tocilizumab Versus Etanercept in Rheumatoid Arthritis: A Randomized Controlled Trial. Arthritis Rheumatol. 2020 Jan;72(1):31-40. doi: 10.1002/art.41095. PMID 31469238

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 3080 patients were enrolled from 353 sites, across 31 countries
Groups:
- Tocilizumab: Participants received 8 mg/kg tocilizumab IV every 4 weeks until switch to another RA therapy or up to 4.9 years.
- Etanercept: Participants received 50 mg etanercept subcutaneously weekly until switch to another RA therapy or up to 4.9 years.
Period: Overall Study
Arm/Group | Tocilizumab | Etanercept
Started | 1538 | 1542
Completed | 1482 | 1475
Not Completed | 56 | 67
Not completed — Death | 30 | 34
Not completed — Lost to Follow-up | 3 | 1
Not completed — Info not recorded | 10 | 16
Not completed — Withdrawal by Subject | 13 | 16

BASELINE CHARACTERISTICS:
Population: Analysis was conducted on the Intention to treat (ITT) population, i.e. all patients randomized who have taken at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tocilizumab | Etanercept | Total
Number analyzed (Participants) | 1538 | 1542 | 3080
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (7.4) | 60.7 (7.6) | 60.7 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1193 | 1202 | 2395
  Male | 345 | 340 | 685

OUTCOME MEASURES:

1. Primary Outcome: Time to First Cardiovascular (CV) Events Adjudication Committee (EAC) (CV-EAC) Adjudicated Event
Description: Prospective comparison of time to first occurrence of any component of the composite of CV death (including events adjudicated as 'Undetermined Cause of Death'), non-fatal myocardial infarction, or non-fatal stroke.
Time Frame: From baseline up to 4.9 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tocilizumab | Etanercept
Number analyzed (Participants) | 1538 | 1542
Months | NA [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to less than 50% of patients experiencing an event | NA [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to less than 50% of patients experiencing an event
Statistical Analysis 1: Comparison: Tocilizumab vs Etanercept; The analysis assessed in the ITT population the hazard ratio of the primary endpoint in TCZ compared to ETA patients. This was done through a comparison of the hazard functions between TCZ and ETA patients. A stratified Cox proportional hazards regression model was used in evaluating the relative CV event rate of TCZ over ETA, with the following randomization factors used as strata: * Previous exposure to anti-TNF (Yes/No) * History of CV events (Yes/No); Test type: Non-Inferiority or Equivalence — In order to reject the null hypothesis and claim non-inferiority of TCZ compared to ETA, a HR point estimate of ≤ 1.278 and upper limit of 95% CI <1.8 was required; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.77 to 1.43]

2. Primary Outcome: Percentage of Patients Reporting a Cardiovascular (CV) Events Adjudication Committee (EAC) (CV-EAC) Adjudicated Event
Description: Percentage of patients reporting any component of the composite of CV death (including events adjudicated as 'Undetermined Cause of Death'), non-fatal myocardial infarction, or non-fatal stroke
Time Frame: From baseline up to 4.9 years
Population: as for baseline characteristics
Measure: Number; unit: Percentage of patients with event
Arm/Group | Tocilizumab | Etanercept
Number analyzed (Participants) | 1538 | 1542
Percentage of patients with event | 5.4 | 5.1

3. Primary Outcome: Time to First CV-EAC Adjudicated Event - Sensitivity Analysis
Description: Prospective comparison of time to first occurrence of any component of the composite of CV death (including events adjudicated as 'Undetermined Cause of Death'), non-fatal myocardial infarction, or non-fatal stroke - Sensitivity Analysis
Time Frame: From Baseline up to 4.9 years
Population: Analyses was conducted on the On-treatment (OT) population, i.e. patients who switched from randomized treatment were censored at the time of treatment switching.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tocilizumab | Etanercept
Number analyzed (Participants) | 1538 | 1542
Months | NA [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to less than 50% of patients experiencing an event | NA [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to less than 50% of patients experiencing an event
Statistical Analysis 1: Comparison: Tocilizumab vs Etanercept; The analysis assessed in the OT population the hazard ratio of the primary endpoint in TCZ compared to ETA patients. This was done through a comparison of the hazard functions between TCZ and ETA patients. A stratified Cox proportional hazards regression model was used in evaluating the relative CV event rate of TCZ over ETA, with the following randomization factors used as strata: * Previous exposure to anti-TNF (Yes/No) * History of CV events (Yes/No); Test type: Non-Inferiority or Equivalence — The non-inferiority margin was only formally tested for the primary ITT analysis'; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.76 to 1.62]

4. Primary Outcome: Percentage of Patients With a CV-EAC Adjudicated Event - Sensitivity Analysis
Description: Percentage of patients with any component of the composite of CV death (including events adjudicated as 'Undetermined Cause of Death'), non-fatal myocardial infarction, or non-fatal stroke - Sensitivity Analysis
Time Frame: From Baseline up to 4.9 years
Population: as for outcome 3
Measure: Number; unit: Percentage of patients with event
Arm/Group | Tocilizumab | Etanercept
Number analyzed (Participants) | 1538 | 1542
Percentage of patients with event | 3.7 | 3.4

5. Primary Outcome: Time to First CV-EAC Adjudicated Event Excluding Undetermined Cause of Death - Sensitivity Analysis
Description: Prospective comparison of time to first occurrence of any component of the composite of CV death (excluding events adjudicated as 'Undetermined Cause of Death'), non-fatal myocardial infarction, or non-fatal stroke - Sensitivity Analyses
Time Frame: From baseline up to 4.9 years
Population: Analysis was conducted on the ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tocilizumab | Etanercept
Number analyzed (Participants) | 1538 | 1542
Months | NA (NA) [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to less than 50% of patients experiencing an event | NA (NA) [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to less than 50% of patients experiencing an event
Statistical Analysis 1: Comparison: Tocilizumab vs Etanercept; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was only formally tested for the primary ITT analysis and not for the sensitivity analysis; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.73 to 1.40]

6. Primary Outcome: Percentage of Patients With a CV-EAC Adjudicated Event Excluding Undetermined Cause of Death - Sensitivity Analysis
Description: Percentage of patients with any component of the composite of CV death (excluding events adjudicated as 'Undetermined Cause of Death'), non-fatal myocardial infarction, or non-fatal stroke - Sensitivity Analyses
Time Frame: From baseline up to 4.9 years
Population: Analysis was conducted on the ITT population
Measure: Number; unit: Percentage of patients with event
Arm/Group | Tocilizumab | Etanercept
Number analyzed (Participants) | 1538 | 1542
Percentage of patients with event | 4.8 | 4.7

7. Primary Outcome: Time to First CV-EAC Adjudicated Event Before Last Direct Contact Date
Description: Prospective comparison of time to first occurrence of any component of the composite of CV death (including events adjudicated as 'Undetermined Cause of Death'), non-fatal myocardial infarction, or non-fatal stroke before last direct contact date (i.e., latest date of visit, IVRS call, or site call).
Time Frame: From Baseline up to 4.9 years
Population: Analysis was conducted on the ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tocilizumab | Etanercept
Number analyzed (Participants) | 1538 | 1542
Months | NA (NA) [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to less than 50% of patients experiencing an event | NA (NA) [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to less than 50% of patients experiencing an event
Statistical Analysis 1: Comparison: Tocilizumab vs Etanercept; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was only formally tested for the primary ITT analysis and not for the sensitivity analysis; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.70 to 1.56]

8. Primary Outcome: Percentage of Participants With a CV-EAC Adjudicated Event Before Last Direct Contact Date
Description: Percentage of participants with any component of the composite of CV death (including events adjudicated as 'Undetermined Cause of Death'), non-fatal myocardial infarction, or non-fatal stroke before last direct contact date (i.e., latest date of visit, IVRS call, or site call).
Time Frame: From Baseline up to 4.9 years
Population: Analysis was conducted on the ITT population
Measure: Number; unit: Percentage of participants with event
Arm/Group | Tocilizumab | Etanercept
Number analyzed (Participants) | 1538 | 1542
Percentage of participants with event | 3.2 | 3.0

9. Secondary Outcome: The Time to First Occurrence of an Expanded CV Composite Endpoint
Description: Prospective comparison of the time to first ccurrence of the expanded composite endpoint. The expanded composite endpoint is defined as the CV composite of the primary endpoint with the addition of non-elective coronary revascularization procedures and hospitalization for unstable angina.
Time Frame: From baseline up to 4.9 years
Population: Analysis was conducted on the ITT population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tocilizumab | Etanercept
Number analyzed (Participants) | 1538 | 1542
Months | NA (NA) [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to less than 50% of patients experiencing an event | NA (NA) [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to less than 50% of patients experiencing an event
Statistical Analysis 1: Comparison: Tocilizumab vs Etanercept; The analysis assessed in the ITT population the hazard ratio of the secondary endpoint in TCZ compared to ETA patients. This was done through a comparison of the hazard functions between TCZ and ETA patients. A stratified Cox proportional hazards regression model was used in evaluating the relative CV event rate of TCZ over ETA, with the following randomization factors used as strata: * Previous exposure to anti-TNF (Yes/No) * History of CV events (Yes/No); Test type: Non-Inferiority or Equivalence — The non-inferiority margin was only formally tested for the primary ITT analysis; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.73 to 1.34]

10. Secondary Outcome: Percentages of Participants With an Expanded CV Composite Endpoint
Description: Percentages of participants with the expanded CV composite endpoint. The expanded composite endpoint is defined as the CV composite of the primary endpoint with the addition of non-elective coronary revascularization procedures and hospitalization for unstable angina.
Time Frame: From baseline up to 4.9 years
Population: Analysis was conducted on the ITT population.
Measure: Number; unit: Percentages of participants
Arm/Group | Tocilizumab | Etanercept
Number analyzed (Participants) | 1538 | 1542
Percentages of participants | 5.5 | 5.4

11. Secondary Outcome: Time to First Occurrence of Individual Component of Primary Endpoint: Non-fatal Myocardial Infarction
Description: Prospective comparison of time to first occurrence of Individual component of primary endpoint: non-fatal Myocardial Infarction
Time Frame: From baseline up to 4.9 years
Population: Anlysis was conducted on the ITT population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tocilizumab | Etanercept
Number analyzed (Participants) | 1538 | 1542
Months | NA (NA) [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to less than 50% of patients experiencing an event | NA (NA) [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to less than 50% of patients experiencing an event
Statistical Analysis 1: Comparison: Tocilizumab vs Etanercept; [analysis description as in outcome 9, analysis 1]; Test type: Non-Inferiority or Equivalence — 'The non-inferiority margin was only formally tested for the primary ITT analysis'; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.54 to 1.49]

12. Secondary Outcome: Percentage of Patients With Individual Component of Primary Endpoint: Non-fatal Myocardial Infarction
Description: Percentage of patients reporting Individual component of primary endpoint: non-fatal Myocardial Infarction
Time Frame: From baseline up to 4.9 years
Population: Anlysis was conducted on the ITT population
Measure: Number; unit: Percentage of patients
Arm/Group | Tocilizumab | Etanercept
Number analyzed (Participants) | 1538 | 1542
Percentage of patients | 1.8 | 2.0

13. Secondary Outcome: Time to First Occurrence of Individual Component of Primary Endpoint: Cardiovascular Death
Description: Prospective comparison of time to first occurrence of Individual component of primary endpoint: cardiovascular death
Time Frame: From baseline up to 4.9 years
Population: Analysis was conducted on the ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tocilizumab | Etanercept
Number analyzed (Participants) | 1538 | 1542
Months | NA (NA) [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to less than 50% of patients experiencing an event | NA (NA) [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to less than 50% of patients experiencing an event
Statistical Analysis 1: Comparison: Tocilizumab vs Etanercept; [analysis description as in outcome 9, analysis 1]; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was only formally tested for the primary ITT analysis; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.64 to 1.63]

14. Secondary Outcome: Percentage of Patients With Individual Component of Primary Endpoint: Cardiovascular Death
Description: Percentage of patients reporting Individual component of primary endpoint: cardiovascular death
Time Frame: From baseline up to 4.9 years
Population: Analysis was conducted on the ITT population
Measure: Number; unit: Percentage of patients
Arm/Group | Tocilizumab | Etanercept
Number analyzed (Participants) | 1538 | 1542
Percentage of patients | 2.3 | 2.3

15. Secondary Outcome: Time to First Occurrence of Individual Component of Primary Endpoint: Non-fatal Stroke
Description: Prospective comparison of time to first occurrence of Individual component of primary endpoint: non-fatal stroke
Time Frame: From baseline up to 4.9 years
Population: Analysis was conducted on the ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tocilizumab | Etanercept
Number analyzed (Participants) | 1538 | 1542
Months | NA (NA) [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to less than 50% of patients experiencing an event | NA (NA) [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to less than 50% of patients experiencing an event
Statistical Analysis 1: Comparison: Tocilizumab vs Etanercept; [analysis description as in outcome 9, analysis 1]; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was only formally tested for the primary ITT analysis; Hazard Ratio (HR) = 1.53, 95% CI 2-sided [0.80 to 2.92]

16. Secondary Outcome: Percentage of Patients With Individual Component of Primary Endpoint: Non-fatal Stroke
Time Frame: From baseline up to 4.9 years
Population: Analysis was conducted on the ITT population
Measure: Number; unit: Percentage of patients
Arm/Group | Tocilizumab | Etanercept
Number analyzed (Participants) | 1538 | 1542
Percentage of patients | 1.6 | 1.0

17. Secondary Outcome: Time to First Occurrence of Individual Component of Primary Endpoint: All-cause Mortality
Description: Prospective comparison of time to first occurrence of Individual component of primary endpoint: All-cause mortality
Time Frame: From baseline up to 4.9 years
Population: Analysis was conducted on the ITT population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tocilizumab | Etanercept
Number analyzed (Participants) | 1538 | 1542
Months | NA (NA) [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to less than 50% of patients experiencing an event | NA (NA) [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to less than 50% of patients experiencing an event
Statistical Analysis 1: Comparison: Tocilizumab vs Etanercept; [analysis description as in outcome 9, analysis 1]; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was only formally tested for the primary ITT analysis; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.70 to 1.41]

18. Secondary Outcome: Percentage of Patients With Individual Component of Primary Endpoint: All-cause Mortality
Description: Percentage of patients reporting Individual component of primary endpoint: All-cause mortality
Time Frame: From baseline up to 4.9 years
Population: Analysis was conducted on the ITT population.
Measure: Number; unit: Percentage of patients
Arm/Group | Tocilizumab | Etanercept
Number analyzed (Participants) | 1538 | 1542
Percentage of patients | 4.2 | 4.2

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the entire course of the study.
Description: Analyses were conducted on the On treatment safety (OTS) population, i.e. all patients randomized who have taken at lease one dose of study medication, with patients censored at time of treatment switch. Patients are presented according to treatment received.
Arm/Group | Etanercept | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 422/1542 | 479/1538
Other Adverse Events (participants affected / at risk) | 910/1542 | 1090/1538
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=1542) | Tocilizumab (N=1538)
ANAEMIA (Blood and lymphatic system disorders) | 9 | 5
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
COAGULOPATHY (Blood and lymphatic system disorders) | 1 | 0
GRANULOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 2 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 4 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 2
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 9 | 7
ADAMS-STOKES SYNDROME (Cardiac disorders) | 1 | 0
ANGINA PECTORIS (Cardiac disorders) | 2 | 8
ANGINA UNSTABLE (Cardiac disorders) | 7 | 4
ATRIAL FIBRILLATION (Cardiac disorders) | 18 | 14
ATRIAL FLUTTER (Cardiac disorders) | 0 | 2
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 2 | 0
BRADYARRHYTHMIA (Cardiac disorders) | 1 | 0
BRADYCARDIA (Cardiac disorders) | 2 | 1
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 4 | 1
CARDIAC FAILURE (Cardiac disorders) | 3 | 11
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 8 | 7
CARDIAC FIBRILLATION (Cardiac disorders) | 0 | 1
CARDIAC TAMPONADE (Cardiac disorders) | 1 | 0
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 0
CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 | 4
CORONARY ARTERY DISEASE (Cardiac disorders) | 3 | 9
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 1 | 1
CORONARY ARTERY STENOSIS (Cardiac disorders) | 2 | 0
HYPERTENSIVE HEART DISEASE (Cardiac disorders) | 0 | 3
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 2 | 0
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 2 | 0
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 | 0
MITRAL VALVE STENOSIS (Cardiac disorders) | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 15 | 10
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 3 | 1
PALPITATIONS (Cardiac disorders) | 1 | 1
POSTINFARCTION ANGINA (Cardiac disorders) | 0 | 1
SILENT MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 0
SINOATRIAL BLOCK (Cardiac disorders) | 1 | 0
SINUS BRADYCARDIA (Cardiac disorders) | 1 | 1
SINUS NODE DYSFUNCTION (Cardiac disorders) | 1 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 1
TACHYCARDIA (Cardiac disorders) | 1 | 1
VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 | 0
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 | 0
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 0 | 1
HYDROCELE (Congenital, familial and genetic disorders) | 1 | 0
DEAFNESS UNILATERAL (Ear and labyrinth disorders) | 1 | 1
VERTIGO (Ear and labyrinth disorders) | 1 | 1
GOITRE (Endocrine disorders) | 1 | 0
HYPERTHYROIDISM (Endocrine disorders) | 0 | 1
HYPOTHYROIDISM (Endocrine disorders) | 0 | 1
CATARACT (Eye disorders) | 2 | 2
CORNEAL PERFORATION (Eye disorders) | 0 | 1
KERATITIS (Eye disorders) | 0 | 1
RETINAL ARTERY OCCLUSION (Eye disorders) | 1 | 1
RETINAL DETACHMENT (Eye disorders) | 1 | 0
SCLERITIS (Eye disorders) | 1 | 0
ULCERATIVE KERATITIS (Eye disorders) | 1 | 2
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 0 | 1
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 2
ACID PEPTIC DISEASE (Gastrointestinal disorders) | 1 | 0
ACUTE ABDOMEN (Gastrointestinal disorders) | 0 | 1
ASCITES (Gastrointestinal disorders) | 0 | 1
COLITIS (Gastrointestinal disorders) | 1 | 1
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 | 0
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 1
CROHN'S DISEASE (Gastrointestinal disorders) | 1 | 0
DIAPHRAGMATIC HERNIA (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 4 | 2
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 1 | 6
DIVERTICULUM (Gastrointestinal disorders) | 0 | 1
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 2 | 1
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 1
DUODENAL ULCER (Gastrointestinal disorders) | 1 | 0
ENTERITIS (Gastrointestinal disorders) | 0 | 1
ENTEROCOLITIS (Gastrointestinal disorders) | 0 | 2
FEMORAL HERNIA (Gastrointestinal disorders) | 0 | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 2
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTRIC ULCER PERFORATION (Gastrointestinal disorders) | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 2 | 4
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 4 | 4
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 1
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 2
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1
INCARCERATED HIATUS HERNIA (Gastrointestinal disorders) | 1 | 0
INCARCERATED UMBILICAL HERNIA (Gastrointestinal disorders) | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 1
LARGE INTESTINAL STENOSIS (Gastrointestinal disorders) | 0 | 1
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 | 4
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 2 | 0
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 0 | 1
MELAENA (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 2
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 1
PALATAL DISORDER (Gastrointestinal disorders) | 1 | 0
PANCREATITIS (Gastrointestinal disorders) | 1 | 4
PANCREATITIS ACUTE (Gastrointestinal disorders) | 3 | 5
PEPTIC ULCER (Gastrointestinal disorders) | 1 | 1
PEPTIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
RETROPERITONEAL FIBROSIS (Gastrointestinal disorders) | 1 | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 2
VOMITING (Gastrointestinal disorders) | 0 | 1
CHEST PAIN (General disorders) | 10 | 3
COMPLICATION ASSOCIATED WITH DEVICE (General disorders) | 0 | 1
DEATH (General disorders) | 4 | 3
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 1
IMPAIRED HEALING (General disorders) | 0 | 1
LOCAL SWELLING (General disorders) | 0 | 1
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 0 | 2
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 5
OEDEMA PERIPHERAL (General disorders) | 1 | 0
PAIN (General disorders) | 0 | 1
PYREXIA (General disorders) | 3 | 3
SUDDEN DEATH (General disorders) | 1 | 3
SWELLING (General disorders) | 0 | 1
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0 | 1
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 3
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 2 | 1
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 6 | 14
HEPATIC VEIN THROMBOSIS (Hepatobiliary disorders) | 1 | 0
HEPATITIS (Hepatobiliary disorders) | 0 | 2
HEPATITIS ACUTE (Hepatobiliary disorders) | 1 | 0
POST CHOLECYSTECTOMY SYNDROME (Hepatobiliary disorders) | 0 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 1
HYPERSENSITIVITY (Immune system disorders) | 0 | 1
OVERLAP SYNDROME (Immune system disorders) | 1 | 0
SARCOIDOSIS (Immune system disorders) | 1 | 0
ABSCESS (Infections and infestations) | 1 | 1
ABSCESS LIMB (Infections and infestations) | 0 | 6
ABSCESS ORAL (Infections and infestations) | 0 | 1
ABSCESS RUPTURE (Infections and infestations) | 1 | 0
ACUTE SINUSITIS (Infections and infestations) | 1 | 0
ANAL ABSCESS (Infections and infestations) | 1 | 0
APPENDICITIS (Infections and infestations) | 0 | 3
ARTHRITIS BACTERIAL (Infections and infestations) | 6 | 9
ARTHRITIS INFECTIVE (Infections and infestations) | 1 | 2
ASPERGILLUS INFECTION (Infections and infestations) | 0 | 1
ATYPICAL PNEUMONIA (Infections and infestations) | 2 | 0
BILIARY SEPSIS (Infections and infestations) | 0 | 1
BRONCHITIS (Infections and infestations) | 4 | 5
BRONCHITIS VIRAL (Infections and infestations) | 1 | 0
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 1 | 0
BURSITIS INFECTIVE (Infections and infestations) | 0 | 2
CELLULITIS (Infections and infestations) | 8 | 24
CELLULITIS STAPHYLOCOCCAL (Infections and infestations) | 1 | 0
CELLULITIS STREPTOCOCCAL (Infections and infestations) | 0 | 1
CERVICITIS (Infections and infestations) | 0 | 1
CHRONIC TONSILLITIS (Infections and infestations) | 0 | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 0
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1 | 0
COLONIC ABSCESS (Infections and infestations) | 0 | 1
DENGUE FEVER (Infections and infestations) | 0 | 1
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 1
DEVICE RELATED SEPSIS (Infections and infestations) | 0 | 1
DISSEMINATED TUBERCULOSIS (Infections and infestations) | 1 | 1
DIVERTICULITIS (Infections and infestations) | 1 | 10
EMPYEMA (Infections and infestations) | 1 | 1
ENDOPHTHALMITIS (Infections and infestations) | 1 | 0
ENTERITIS INFECTIOUS (Infections and infestations) | 2 | 0
EPIDIDYMITIS (Infections and infestations) | 1 | 1
EPIGLOTTITIS (Infections and infestations) | 0 | 2
ERYSIPELAS (Infections and infestations) | 2 | 11
ESCHERICHIA PYELONEPHRITIS (Infections and infestations) | 0 | 1
ESCHERICHIA SEPSIS (Infections and infestations) | 0 | 1
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
FUNGAL SKIN INFECTION (Infections and infestations) | 0 | 1
GASTROENTERITIS (Infections and infestations) | 6 | 3
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 0 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 1
GROIN ABSCESS (Infections and infestations) | 1 | 0
HAEMATOMA INFECTION (Infections and infestations) | 0 | 1
HAEMOPHILUS SEPSIS (Infections and infestations) | 0 | 1
HERPANGINA (Infections and infestations) | 0 | 1
HERPES ZOSTER (Infections and infestations) | 4 | 2
INFECTED DERMAL CYST (Infections and infestations) | 1 | 1
INFECTION (Infections and infestations) | 1 | 0
INFECTIOUS COLITIS (Infections and infestations) | 2 | 0
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 1 | 3
INFECTIVE ANEURYSM (Infections and infestations) | 0 | 1
INFLUENZA (Infections and infestations) | 1 | 1
INJECTION SITE ABSCESS (Infections and infestations) | 0 | 1
INTERVERTEBRAL DISCITIS (Infections and infestations) | 0 | 1
LOCALISED INFECTION (Infections and infestations) | 0 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1
LUDWIG ANGINA (Infections and infestations) | 0 | 1
LUNG ABSCESS (Infections and infestations) | 0 | 1
LUNG INFECTION (Infections and infestations) | 1 | 0
LUNG INFECTION PSEUDOMONAL (Infections and infestations) | 0 | 1
MASTOIDITIS (Infections and infestations) | 0 | 1
MENINGITIS (Infections and infestations) | 0 | 2
MUSCLE ABSCESS (Infections and infestations) | 1 | 1
NASAL ABSCESS (Infections and infestations) | 1 | 0
NEUROSYPHILIS (Infections and infestations) | 0 | 1
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 2 | 0
OPHTHALMIC HERPES SIMPLEX (Infections and infestations) | 1 | 0
OPHTHALMIC HERPES ZOSTER (Infections and infestations) | 1 | 2
OSTEOMYELITIS (Infections and infestations) | 2 | 2
OSTEOMYELITIS CHRONIC (Infections and infestations) | 1 | 0
OTITIS EXTERNA (Infections and infestations) | 0 | 1
PAPILLOMA VIRAL INFECTION (Infections and infestations) | 0 | 1
PERIHEPATIC ABSCESS (Infections and infestations) | 1 | 0
PERITONITIS (Infections and infestations) | 0 | 3
PERITONSILLAR ABSCESS (Infections and infestations) | 1 | 0
PHARYNGITIS (Infections and infestations) | 1 | 0
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 41 | 47
PNEUMONIA BACTERIAL (Infections and infestations) | 1 | 1
PNEUMONIA INFLUENZAL (Infections and infestations) | 1 | 0
PNEUMONIA MYCOPLASMAL (Infections and infestations) | 1 | 0
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 0 | 1
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 1 | 0
PNEUMONIA VIRAL (Infections and infestations) | 1 | 0
POST PROCEDURAL INFECTION (Infections and infestations) | 0 | 2
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 4 | 1
PSEUDOMONAS INFECTION (Infections and infestations) | 0 | 1
PULMONARY TUBERCULOMA (Infections and infestations) | 1 | 0
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 | 1
PYELONEPHRITIS (Infections and infestations) | 1 | 5
RECTAL ABSCESS (Infections and infestations) | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 2
SALPINGITIS (Infections and infestations) | 0 | 1
SCROTAL ABSCESS (Infections and infestations) | 0 | 1
SEPSIS (Infections and infestations) | 7 | 6
SEPTIC SHOCK (Infections and infestations) | 3 | 3
SINUSITIS (Infections and infestations) | 2 | 0
SOFT TISSUE INFECTION (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 1
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 | 2
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 1 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 3 | 2
TONGUE ABSCESS (Infections and infestations) | 1 | 0
TONSILLITIS (Infections and infestations) | 0 | 1
TOXIC SHOCK SYNDROME STREPTOCOCCAL (Infections and infestations) | 0 | 1
TRACHEITIS (Infections and infestations) | 1 | 0
TUBERCULOSIS (Infections and infestations) | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1
URINARY TRACT INFECTION (Infections and infestations) | 12 | 7
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 | 1
UROSEPSIS (Infections and infestations) | 2 | 1
VIRAL INFECTION (Infections and infestations) | 0 | 1
VIRAL PHARYNGITIS (Infections and infestations) | 1 | 0
WEST NILE VIRAL INFECTION (Infections and infestations) | 1 | 0
WOUND INFECTION (Infections and infestations) | 1 | 1
ACCIDENT AT WORK (Injury, poisoning and procedural complications) | 0 | 1
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
ARTHROPOD STING (Injury, poisoning and procedural complications) | 1 | 0
COMMINUTED FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
CONTUSION (Injury, poisoning and procedural complications) | 1 | 1
DISLOCATION OF VERTEBRA (Injury, poisoning and procedural complications) | 2 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 2
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 3 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 6 | 5
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FRACTURE DISPLACEMENT (Injury, poisoning and procedural complications) | 1 | 0
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 1 | 0
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 12 | 4
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 4 | 3
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 | 2
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 2 | 3
JOINT INJURY (Injury, poisoning and procedural complications) | 1 | 0
LIGAMENT INJURY (Injury, poisoning and procedural complications) | 1 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
PNEUMOTHORAX TRAUMATIC (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL FISTULA (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 2
RESPIRATORY FUME INHALATION DISORDER (Injury, poisoning and procedural complications) | 0 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 4 | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
STOMAL HERNIA (Injury, poisoning and procedural complications) | 0 | 1
STRESS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
SUBCUTANEOUS HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 2
SYNOVIAL RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 2 | 1
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
ULNA FRACTURE (Injury, poisoning and procedural complications) | 1 | 2
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 2
WOUND (Injury, poisoning and procedural complications) | 0 | 1
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 1
WRIST FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
EOSINOPHIL COUNT INCREASED (Investigations) | 1 | 0
HAEMATOCRIT ABNORMAL (Investigations) | 0 | 1
HAEMOGLOBIN ABNORMAL (Investigations) | 0 | 1
LIVER FUNCTION TEST INCREASED (Investigations) | 1 | 0
STAPHYLOCOCCUS TEST POSITIVE (Investigations) | 1 | 0
SYNOVIAL FLUID WHITE BLOOD CELLS POSITIVE (Investigations) | 0 | 1
TRANSAMINASES INCREASED (Investigations) | 1 | 0
TROPONIN INCREASED (Investigations) | 2 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 4 | 5
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
DIABETIC COMPLICATION (Metabolism and nutrition disorders) | 1 | 0
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 3 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 3 | 1
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 | 0
BURSITIS (Musculoskeletal and connective tissue disorders) | 2 | 2
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
FASCIITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
FINGER DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 | 1
FISTULA (Musculoskeletal and connective tissue disorders) | 0 | 1
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 3 | 2
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 3
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 6 | 5
KNEE DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 | 1
LIMB DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 | 0
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
MORPHOEA (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 22 | 14
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 4 | 2
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 2 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 1
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 15 | 12
RHEUMATOID NODULE (Musculoskeletal and connective tissue disorders) | 0 | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 1 | 0
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 | 1
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 | 1
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
ANAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
BENIGN ANORECTAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BENIGN NEOPLASM OF CERVIX UTERI (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
CARCINOID TUMOUR OF THE GASTROINTESTINAL TRACT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CARCINOID TUMOUR PULMONARY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CARDIAC MYXOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CENTRAL NERVOUS SYSTEM LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CEREBRAL HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CHOLANGIOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ENDOMETRIAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
GLIOBLASTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
INTESTINAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
INTRADUCTAL PROLIFERATIVE BREAST LESION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
LUNG ADENOCARCINOMA STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
MALIGNANT MELANOMA STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MARJOLIN'S ULCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTATIC GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OVARIAN ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PARAPROTEINAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PHARYNGEAL NEOPLASM BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PITUITARY TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PLASMA CELL MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA OF LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA OF THE TONGUE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SQUAMOUS ENDOMETRIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
THYROID ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
TONGUE NEOPLASM MALIGNANT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
TUMOUR INVASION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
AMYOTROPHIC LATERAL SCLEROSIS (Nervous system disorders) | 1 | 0
BALANCE DISORDER (Nervous system disorders) | 1 | 0
BRAIN STEM INFARCTION (Nervous system disorders) | 0 | 1
CAROTID ARTERY DISEASE (Nervous system disorders) | 1 | 0
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 | 1
CEREBRAL HAEMATOMA (Nervous system disorders) | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 2 | 1
CEREBRAL ISCHAEMIA (Nervous system disorders) | 2 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 8 | 14
CEREBROVASCULAR DISORDER (Nervous system disorders) | 1 | 1
CERVICAL CORD COMPRESSION (Nervous system disorders) | 0 | 1
CERVICAL RADICULOPATHY (Nervous system disorders) | 1 | 0
COMA (Nervous system disorders) | 1 | 0
DEMENTIA (Nervous system disorders) | 0 | 1
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 0 | 1
DIABETIC COMA (Nervous system disorders) | 0 | 1
DYSARTHRIA (Nervous system disorders) | 0 | 1
DYSKINESIA (Nervous system disorders) | 0 | 1
EMBOLIC STROKE (Nervous system disorders) | 1 | 0
ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
EPILEPSY (Nervous system disorders) | 0 | 3
FACIAL PARALYSIS (Nervous system disorders) | 0 | 1
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 0 | 1
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 | 0
HEMIPARESIS (Nervous system disorders) | 1 | 0
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
HYPERTENSIVE ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
INTRACRANIAL ANEURYSM (Nervous system disorders) | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 5 | 5
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
LUMBAR RADICULOPATHY (Nervous system disorders) | 2 | 0
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
MIGRAINE (Nervous system disorders) | 0 | 1
MYASTHENIA GRAVIS (Nervous system disorders) | 1 | 0
PARAESTHESIA (Nervous system disorders) | 1 | 1
PARKINSON'S DISEASE (Nervous system disorders) | 1 | 0
PRESYNCOPE (Nervous system disorders) | 2 | 0
REVERSIBLE ISCHAEMIC NEUROLOGICAL DEFICIT (Nervous system disorders) | 1 | 0
RUPTURED CEREBRAL ANEURYSM (Nervous system disorders) | 0 | 1
SCIATICA (Nervous system disorders) | 3 | 1
SEIZURE (Nervous system disorders) | 1 | 1
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 | 2
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 3 | 1
SYNCOPE (Nervous system disorders) | 1 | 0
TRANSIENT GLOBAL AMNESIA (Nervous system disorders) | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 3 | 9
VASCULAR DEMENTIA (Nervous system disorders) | 0 | 1
DEVICE BREAKAGE (Product Issues) | 1 | 0
DEVICE DISLOCATION (Product Issues) | 0 | 3
DEVICE FAILURE (Product Issues) | 0 | 1
DEVICE LOOSENING (Product Issues) | 0 | 1
BURNOUT SYNDROME (Psychiatric disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 1
DELIRIUM (Psychiatric disorders) | 0 | 1
DELIRIUM TREMENS (Psychiatric disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 2 | 0
MAJOR DEPRESSION (Psychiatric disorders) | 0 | 1
MENTAL DISORDER (Psychiatric disorders) | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 1
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 | 1
SCHIZOAFFECTIVE DISORDER BIPOLAR TYPE (Psychiatric disorders) | 0 | 1
SUICIDAL IDEATION (Psychiatric disorders) | 0 | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 5 | 3
CALCULUS BLADDER (Renal and urinary disorders) | 0 | 1
CALCULUS URINARY (Renal and urinary disorders) | 2 | 1
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 | 1
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 1 | 0
END STAGE RENAL DISEASE (Renal and urinary disorders) | 1 | 0
GLOMERULONEPHRITIS CHRONIC (Renal and urinary disorders) | 0 | 1
HYDRONEPHROSIS (Renal and urinary disorders) | 1 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 3 | 3
OBSTRUCTIVE NEPHROPATHY (Renal and urinary disorders) | 0 | 1
PELVI-URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 | 1
RENAL COLIC (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 3 | 2
TUBULOINTERSTITIAL NEPHRITIS (Renal and urinary disorders) | 1 | 0
URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 | 1
URETEROLITHIASIS (Renal and urinary disorders) | 1 | 2
URETHRAL STENOSIS (Renal and urinary disorders) | 0 | 1
URINARY RETENTION (Renal and urinary disorders) | 0 | 1
ACQUIRED PHIMOSIS (Reproductive system and breast disorders) | 1 | 0
BREAST FIBROSIS (Reproductive system and breast disorders) | 1 | 0
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 0 | 1
CERVICAL POLYP (Reproductive system and breast disorders) | 0 | 1
CYSTOCELE (Reproductive system and breast disorders) | 0 | 2
GENITAL PROLAPSE (Reproductive system and breast disorders) | 0 | 1
METRORRHAGIA (Reproductive system and breast disorders) | 0 | 1
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 0
OVARIAN CYST TORSION (Reproductive system and breast disorders) | 0 | 1
RECTOCELE (Reproductive system and breast disorders) | 1 | 0
SPERMATOCELE (Reproductive system and breast disorders) | 0 | 1
UTERINE POLYP (Reproductive system and breast disorders) | 1 | 0
UTERINE PROLAPSE (Reproductive system and breast disorders) | 1 | 1
VAGINAL HAEMATOMA (Reproductive system and breast disorders) | 0 | 1
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ALVEOLITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 5 | 2
ASTHMATIC CRISIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
BRONCHIAL HYPERREACTIVITY (Respiratory, thoracic and mediastinal disorders) | 0 | 1
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 0 | 1
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
BRONCHOSTENOSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 7 | 10
CHRONIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 | 5
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYDROTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 3 | 5
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 5 | 6
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 11 | 1
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PULMONARY GRANULOMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY SARCOIDOSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 2 | 1
BLISTER (Skin and subcutaneous tissue disorders) | 0 | 1
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 | 0
DERMAL CYST (Skin and subcutaneous tissue disorders) | 1 | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 1 | 0
HYPERSENSITIVITY VASCULITIS (Skin and subcutaneous tissue disorders) | 1 | 0
PEMPHIGOID (Skin and subcutaneous tissue disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 1
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN NECROSIS (Skin and subcutaneous tissue disorders) | 0 | 2
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 4
URTICARIA (Skin and subcutaneous tissue disorders) | 2 | 0
VASCULITIC ULCER (Skin and subcutaneous tissue disorders) | 0 | 1
ABDOMINAL HERNIA REPAIR (Surgical and medical procedures) | 1 | 0
ANAL FISTULA EXCISION (Surgical and medical procedures) | 1 | 0
ANGIOPLASTY (Surgical and medical procedures) | 0 | 1
APPENDICECTOMY (Surgical and medical procedures) | 0 | 1
CARDIAC PACEMAKER REPLACEMENT (Surgical and medical procedures) | 0 | 1
COLOSTOMY CLOSURE (Surgical and medical procedures) | 1 | 0
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 | 1
IMPLANTABLE DEFIBRILLATOR INSERTION (Surgical and medical procedures) | 1 | 0
KNEE ARTHROPLASTY (Surgical and medical procedures) | 0 | 1
LARGE INTESTINE ANASTOMOSIS (Surgical and medical procedures) | 0 | 1
MITRAL VALVE REPLACEMENT (Surgical and medical procedures) | 1 | 0
SEQUESTRECTOMY (Surgical and medical procedures) | 0 | 1
UMBILICAL HERNIA REPAIR (Surgical and medical procedures) | 0 | 1
AORTIC ANEURYSM (Vascular disorders) | 4 | 3
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 0 | 1
AORTIC CALCIFICATION (Vascular disorders) | 0 | 1
AORTIC DISSECTION (Vascular disorders) | 1 | 1
AORTIC STENOSIS (Vascular disorders) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 8 | 6
EMBOLISM ARTERIAL (Vascular disorders) | 1 | 0
FEMORAL ARTERY EMBOLISM (Vascular disorders) | 1 | 0
HAEMATOMA (Vascular disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 6 | 4
HYPERTENSIVE CRISIS (Vascular disorders) | 2 | 1
HYPERTENSIVE EMERGENCY (Vascular disorders) | 1 | 0
HYPOTENSION (Vascular disorders) | 1 | 2
INFARCTION (Vascular disorders) | 1 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 2 | 1
PERIPHERAL ISCHAEMIA (Vascular disorders) | 2 | 3
PERIPHERAL VENOUS DISEASE (Vascular disorders) | 1 | 2
RHEUMATOID VASCULITIS (Vascular disorders) | 1 | 0
SUBCLAVIAN ARTERY OCCLUSION (Vascular disorders) | 1 | 0
THROMBOSIS (Vascular disorders) | 1 | 2
VARICOSE VEIN (Vascular disorders) | 0 | 1
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 3 | 1
MANIA (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=1542) | Tocilizumab (N=1538)
LEUKOPENIA (Blood and lymphatic system disorders) | 21 | 85
NEUTROPENIA (Blood and lymphatic system disorders) | 33 | 92
DIARRHOEA (Gastrointestinal disorders) | 84 | 140
BRONCHITIS (Infections and infestations) | 185 | 244
NASOPHARYNGITIS (Infections and infestations) | 141 | 239
PHARYNGITIS (Infections and infestations) | 76 | 113
SINUSITIS (Infections and infestations) | 78 | 88
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 193 | 243
URINARY TRACT INFECTION (Infections and infestations) | 150 | 174
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 44 | 120
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 52 | 143
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 106 | 143
BACK PAIN (Musculoskeletal and connective tissue disorders) | 92 | 147
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 132 | 152
HEADACHE (Nervous system disorders) | 68 | 103
COUGH (Respiratory, thoracic and mediastinal disorders) | 76 | 127
HYPERTENSION (Vascular disorders) | 158 | 200

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.